CLINICAL TRIAL: NCT07406451
Title: Inspiratory Muscle Training Enhances Jumping Power and Shoot-ing Performance in Elite Air Pistol Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gümüşhane Universıty (Other)
Responsible Party: Principal Investigator, Coşkun YILMAZ, director, Gümüşhane Universıty
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025-019
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Inspiratory Muscle Training; Shooting Performance; Jump Performance; Precision Sport Performance
Keywords: Inspiratory Muscle Training; Jump performance; Shooting performance; SCATT; Reaction Time
MeSH Terms: interventions — Population Groups; Control Groups

STUDY DESIGN:
Intervention Model Description: Participants performed inspiratory muscle training using a POWERbreathe® Classic device. Training consisted of two daily sessions of 30 resisted breaths, six days per week, for four weeks. Initial resistance was set at 40% of maximal inspiratory pressure (MIP) and progressively increased weekly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory Muscle Training (IMT) Group (Experimental): Participants performed inspiratory muscle training using a POWERbreathe® Classic device. Training consisted of two daily sessions of 30 resisted breaths, six days per week, for four weeks. Initial resistance was set at 40% of maximal inspiratory pressure (MIP) and progressively increased weekly.
  Interventions: Other: Inspiratory Muscle Training (IMT) Group; Other: Control Group (A):
- Control Group (No Intervention): Participants continued their regular air pistol training routines without inspiratory muscle training.

INTERVENTIONS:
Other: Inspiratory Muscle Training (IMT) Group — Participants performed inspiratory muscle training using a POWERbreathe® Classic device. Training consisted of two daily sessions of 30 resisted breaths, six days per week, for four weeks. Initial resistance was set at 40% of maximal inspiratory pressure (MIP) and progressively increased weekly.
  Arms: Inspiratory Muscle Training (IMT) Group
Other: Control Group (A): — Participants continued their regular air pistol training routines without inspiratory muscle training.
  Arms: Inspiratory Muscle Training (IMT) Group

SUMMARY:
This randomized controlled trial investigated the effects of a four-week inspiratory muscle training (IMT) program on physical and motor performance parameters and shooting accuracy in elite male air pistol athletes. Twenty athletes were randomly assigned to either an IMT group or a control group. Outcome measures included jumping performance, reaction time, flexibility, and shooting accuracy assessed via the SCATT system. The findings demonstrated that IMT significantly improved lower-limb explosive power and shooting performance without affecting reaction time or flexibility.

DETAILED DESCRIPTION:
Air pistol shooting is a precision sport requiring postural stability, neuromuscular coordination, and controlled breathing. Inspiratory muscle training has been shown to enhance respiratory muscle strength, trunk stability, and neuromuscular efficiency. However, evidence regarding its effects in precision sports is limited.

This study employed a four-week parallel-group randomized controlled design to examine whether IMT improves jumping performance, reaction time, and shooting accuracy in elite air pistol athletes. The IMT group performed twice-daily resisted breathing sessions using a POWERbreathe® device, while the control group continued standard training. Performance outcomes were assessed before and after the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Male athletes aged 18-35 years
* Minimum of 3 years of systematic air pistol shooting experience
* Regular training for at least the previous 6 months
* Medically cleared for physical activity

Exclusion Criteria:

* History of respiratory, cardiovascular, neurological, or musculoskeletal disorders
* Current injury affecting performance
* Participation in respiratory muscle training within the last 6 months

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male athletes aged 18-35 years
Enrollment: 20 (Actual)
Dates: Start 2025-09-05 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Shooting Performance (SCATT Score) | 4 weeks
  Shooting accuracy and stability assessed using the SCATT shooting simulation system

SECONDARY OUTCOMES:
Countermovement Jump Height and Power | 4 Weeks
  Measured using OptoJump Next system
Squat Jump Height and Power | 4 Weeks
  Measured using OptoJump Next system
Visual Reaction Time | 4 weeks
  Assessed using Cognitech reaction time tester
Auditory Reaction Time | 4 week
  Assessed using Cognitech reaction time tester
Flexibility (Sit-and-Reach Test) | 4 week
  Flexibility (Sit-and-Reach Test)

CONTACTS AND LOCATIONS:
Locations (1):
- Gumushane Univetsity, Gümüşhane, Trabzon, Ordu, Giresun, Rize, Artvin, Gümüşhane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data collected in this study will not be shared with other researchers due to the need to protect participant confidentiality and the lack of permission for data sharing within the scope of informed consent.